CLINICAL TRIAL: NCT02456766
Title: A Multicenter Clinical Study on the Comparison of Acoustic Attenuation Parameter Using FibroTouch With Liver Biopsy for the Diagnosis of Hepatic Steatosis
Brief Title: Comparison of Acoustic Attenuation Parameter Using FibroTouch With Liver Biopsy for Diagnosis of Hepatic Steatosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuxi Hisky Medical Technology Co Ltd (Industry)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Guangzhou First People's Hospital (Other); Ruijin Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); No.85 Hospital, Changning, Shanghai, China (Other); The Second Hospital of Nanjing Medical University (Other); Sichuan Academy of Medical Sciences (Other); Second People's Hospital of Hangzhou (Unknown)
Responsible Party: Sponsor
Other Study IDs: TG1310FT
Record Dates: First submitted 2015-03-22; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Fatty Liver; Hepatic Steatosis; Liver Steatosis
Keywords: FibroTouch; acoustic attenuation parameter; liver biopsy; hepatic steatosis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Liver Biospy Specimens

GROUPS / COHORTS (4):
- F0: Liver Steatosis Grade: <5%
  Interventions: Device: FibroTouch; Procedure: Liver Biopsy
- F1: Liver Steatosis Grade: 5-33%
  Interventions: Device: FibroTouch; Procedure: Liver Biopsy
- F2: Liver Steatosis Grade: 34-66%
  Interventions: Device: FibroTouch; Procedure: Liver Biopsy
- F3: Liver Steatosis Grade: > 66%
  Interventions: Device: FibroTouch; Procedure: Liver Biopsy

INTERVENTIONS:
Device: FibroTouch
Procedure: Liver Biopsy

SUMMARY:
This will be a multi-center, prospective, controlled study. It is expected that about 240 subjects from 10 study centers will be enrolled, and 224 effective subjects will be statistically analyzed in the end, in which 56 effective subjects with stage F0 (25%), 56 effective subjects with stage F1 (25%), 56 effective subjects with stage F2 (25%), 56 effective subjects with stage F3 (25%). By comparison of the result of FibroTouch examination with that of liver biopsy, their specificities, sensitivities and accuracies for diagnosis of liver steatosis will be identified.

The patients with liver diseases who need to have a liver biopsy in hospital and meet all of the inclusion criteria and none of the exclusion criteria, may participate in this study. Within two weeks of FibroTouch examination, subjects are required to have qualified histological specimens of liver biopsy for comparation.

ELIGIBILITY:
Inclusion Criteria:

* Subject at the age of 18 to 65 years, non-limited gender.
* Within two weeks of FibroTouch examination, qualified histological specimens of liver biopsy are required. Using the liver biopsy needle of 16G or 14CT, puncture and remove more than 2.0 centimeters long liver tissue (including at least 11 portal areas, no less than 6 complete portal areas and the minimum length of specimen should be more than 1.0 centimeter).
* Willing and able to abide by all principles and complete all study procedures.
* Willing and can provide written informed consent form by patient or patient's legal guardian.

Exclusion Criteria:

* Subject with active or suspected cancer or history of malignant tumor by evidence within 5 years before enrolling. And the subject who has the liver malignant tumors injury cannot participate in this study.
* There is evidence that the subject has a history of alcohol overdoses* or drug abuse. Definition of alcohol overdoses: 40 gram (g)/day for male and 40 g/day for female. Alcohol intake (g) = the volume of drinking (ml) × alcohol percentage (%, v/v) × 0.8 (g/ml); 1g alcohol is the equal of 25-40 ml of beer, 8-10ml of Chinese rice wine, 5-12ml of (grape) wine, 3-7ml of health care liquor or Chinese spirits.
* Subject with alcoholic liver disease and hepatitis C.
* Pregnant or nursing woman, and subject with a pregnant plan and is unwilling to take contraceptive measures during this study.
* Subject with history of organ transplantation or has functional grafts (except for the cornea or hair graft).
* Subject with non-healing wound on the right upper abdomen at this moment.
* In the investigator's opinion, the subject is unsuitable to participate in the study as he or she has a history of serious illness, or other evidence shown that the subject has any other serious illness.
* Subject who participates in other clinical trial at the same time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects with liver diseases who need to have a liver biopsy in hospital and meet all of the inclusion criteria and none of the exclusion criteria, may participate in this study. Within two weeks of FibroTouch examination, subjects are required to have qualified histological specimens of liver biopsy for comparation.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The coincidence for diagnosis of hepatic steatosis between fat attenuation parameter (FAP) of FibroTouch and liver biopsy by ROC analysis | Within two weeks of FibroTouch examination
  Performance of fat attenuation parameter (FAP, dB/m) of FibroTouch will be assessed using ROC analysis for the detection of hepatic steatosis stage F0 (<5%), stage F1 (5%-33%), stage F2 (34%-66%), and stage F3 (2>66%) using liver biopsy as the reference.

CONTACTS AND LOCATIONS:
Overall Officials: Lungen LU, MD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (8):
- China (8):
  - Sichuan Academy of Medical Sciences &Sichuan Provincial People's Hospital, Chengdu
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Second People's Hospital of Hangzhou, Hangzhou
  - The Second Hospital Of Nanjing, Nanjing
  - Ruijin Hospital, Shanghai
  - Shanghai 85 Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

REFERENCES:
- [Derived] Qu Y, Song YY, Chen CW, Fu QC, Shi JP, Xu Y, Xie Q, Yang YF, Zhou YJ, Li LP, Xu MY, Cai XB, Zhang QD, Yu H, Fan JG, Lu LG. Diagnostic Performance of FibroTouch Ultrasound Attenuation Parameter and Liver Stiffness Measurement in Assessing Hepatic Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease. Clin Transl Gastroenterol. 2021 Apr 13;12(4):e00323. doi: 10.14309/ctg.0000000000000323. PMID 33848277